CLINICAL TRIAL: NCT05918406
Title: A Phase 4, Single Center, Open Label Study Evaluating the Safety of the Nasal Guide Utilized During Administration With Tyrvaya
Brief Title: Phase 4 Study Evaluating the Safety of the Nasal Guide With Tyrvaya
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPP-009
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye; Keratoconjunctivitis Sicca
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca

STUDY DESIGN:
Intervention Model Description: Nasal guide will be used to aid in the administration of Tyrvaya® (varenicline solution 0.03 mg) Nasal Spray
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nasal Guide (Experimental): Use of Nasal Guide with administration of Tyrvaya (varenicline solution 0.03 mg) BID
  Interventions: Combination Product: Nasal Guide

INTERVENTIONS:
Combination Product: Nasal Guide — Use of Nasal Guide with administration of Tyrvaya (varenicline solution 0.03 mg) BID

SUMMARY:
The objective of this study is to determine the safety of the nasal guide when utilized to aid in the administration of Tyrvaya (varenicline solution 0.03mg) Nasal Spray

DETAILED DESCRIPTION:
Protocol OPP-009 is a single center, open-label study to evaluate the safety of the nasal guide during administration of Tyrvaya (varenicline solution 0.03mg) Nasal Spray. Approximately 30 subjects at least 18 years of age will be enrolled at one clinical study site and will receive the nasal guide for use with the administration of Tyrvaya for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age
2. Have provided verbal and written informed consent
3. Willing to comply with all study related visits and procedures

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2023-08-18 (Actual); Study Completion 2023-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marian Macsai, MD, Study Director — Oyster Point Pharma
Locations (2):
- United States (2):
  - United States, New Jersey, Edison, New Jersey
  - United States, New Jersey, Woodland Park, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Tyrvaya (Varenicline Solution 0.3mg) Nasal Spray Administered With the Nasal Guide: Subjects will administer Tyrvaya BID with nasal guide for 7 days
Period: Overall Study
Arm/Group | Tyrvaya (Varenicline Solution 0.3mg) Nasal Spray Administered With the Nasal Guide
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nasal Guide
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (18.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events with use of the nasal guide
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Tyrvaya Nasal Spray Administered With the Nasal Guide: Subjects will administer Tyrvaya (varenicline solution 0.3mg) BID with nasal guide for 7 days
Arm/Group | Tyrvaya Nasal Spray Administered With the Nasal Guide
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: AE collection will start following the first administration of Tyrvaya® utilizing the nasal guide until the last follow up visit of the study at 7 days.
Description: The safety population will include all enrolled subjects who received at least one Tyrvaya® administered with the nasal guide.
Arm/Group | Tyrvaya (Varenicline Solution 0.3mg) Nasal Spray Administered With the Nasal Guide
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tyrvaya (Varenicline Solution 0.3mg) Nasal Spray Administered With the Nasal Guide (N=30)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT05918406/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT05918406/SAP_001.pdf